CLINICAL TRIAL: NCT05526729
Title: Special Drug Use Observational Study With Beovu Kit for Intravitreal Injection (DME, CRTH258B1401)
Brief Title: Special Drug Use Observational Study With Beovu Kit for Intravitreal Injection
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRTH258B1401
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Macular Edema
Keywords: diabetic macular edema; DME; NIS; Japan; PMS; Beovu
MeSH Terms: interventions — brolucizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Beovu: Patients prescribed with Beovu for diabetic macular edema
  Interventions: Other: Beovu

INTERVENTIONS:
Other: Beovu — Prospective observational study. There was no treatment allocation. Patients prescribed with Beovu for the first time for diabetic macular edema were eligible to enroll into this study.
  Other Names: Brolucizumab

SUMMARY:
This was a primary data collection-based observational special drug-use surveillance to be conducted in accordance with the Good Post-marketing Study Practice (GPSP) ordinance.

DETAILED DESCRIPTION:
This study aimed to evaluate the safety of Beovu kit for intravitreal injection in clinical use in diabetic macular edema (DME) patients.

The observation period was 1 year (52 weeks) from the first Beovu administration in the primary treated eye.

In patients discontinuing treatment with Beovu in the primary treated eye before Week 52, the following observation periods applied.

* Date of last Beovu dose + 90 days* in primary treated eye > Week 52: up to Week 52
* Date of last Beovu dose + 90 days* in primary treated eye ≤ Week 52: up to last dosing date in the primary treated eye + 90 days *90 days: to collect as much data as possible considering clinical effects

ELIGIBILITY:
Inclusion Criteria:

1. Patients must provide written consent to cooperate in this study before the start of treatment with Beovu
2. Patients using Beovu for the first time for the following indication • Indication: diabetic macular edema

Exclusion Criteria:

1. Patients with a history of treatment with a drug containing the same ingredient (brolucizumab) as Beovu

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients using Beovu for the first time for diabetic macular edema in Japan
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with adverse events corresponding to each of the safety specifications during the observation period | Up to 52 weeks
  Proportion of patients with adverse events corresponding to each of the safety specifications during the observation period was collected.
  Safety specifications: intraocular inflammation, endophthalmitis, intraocular pressure elevation, retinal detachment and retinal tear, retinal arterial embolic events, non-ocular arterial thromboembolic events, retinal vasculitis and retinal vascular occlusion
Proportions of patients with adverse events in the eyes on therapy during the observation period | Up to 52 weeks
  Proportions of patients with adverse events in the eyes on therapy during the observation period was collected
Proportion of patients with systemic adverse events during the observation period | Up to 52 weeks
  Proportion of patients with systemic (non-ocular) adverse events during the observation period was collected

SECONDARY OUTCOMES:
Proportion of patients with serious adverse events (SAEs) and adverse reactions in the eyes on therapy during the observation period | Up to 52 weeks
  Proportion of patients with serious adverse events (SAEs) and adverse reactions in the eyes on therapy during the observation period was collected
Proportion of patients with systemic SAEs and adverse reactions during the observation period | Up to 52 weeks
  Proportion of patients with systemic (non-ocular) SAEs and adverse reactions during the observation period was collected
Proportion of patients with SAEs, adverse reactions and serious adverse reactions corresponding to the safety specifications during the observation period | Up to 52 weeks
  Proportion of patients with SAEs, adverse reactions and serious adverse reactions corresponding to the safety specifications during the observation period was collected.
  Safety specifications: intraocular inflammation, endophthalmitis, intraocular pressure elevation, retinal detachment and retinal tear, retinal arterial embolic events, non-ocular arterial thromboembolic events, retinal vasculitis and retinal vascular occlusion
Incidences of adverse events by risk factor of the safety specifications | Up to 52 weeks
  Incidences of adverse events by risk factor of the safety specifications (primary treated eyes only) was collected.
  Safety specifications: intraocular inflammation, endophthalmitis, intraocular pressure elevation, retinal detachment and retinal tear, retinal arterial embolic events, non-ocular arterial thromboembolic events, retinal vasculitis and retinal vascular occlusion
Proportion of patients with VA worsening during the observation period | Up to 52 weeks
  Proportion of patients with decimal VA worsening during the observation period was calculated.
  VA was measured in best corrected visual acuity (BCVA). BCVA is the best possible vision that an eye can achieve with the use of glasses or contact lenses
Proportion of patients by administration status in the induction and maintenance phase during the observation period | Up to 52 weeks
  Number of patients by administration status (yes/no) in the induction and maintenance phase during the observation period was collected
Proportion of patients by treated eye in the induction and maintenance phase during the observation period | Up to 52 weeks
  Number of patients by treated eye (right eye/left eye) in the induction and maintenance phase during the observation period was collected

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (64):
- Japan (64):
  - Novartis Investigative Site, Nagakute, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Kisarazu, Chiba
  - Novartis Investigative Site, Urayasu, Chiba
  - Novartis Investigative Site, Yoshida-gun, Fukui
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Fukushima, Fukushima
  - Novartis Investigative Site, Mizunami, Gifu
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Asahikawa, Hokkaido
  - Novartis Investigative Site, Hakodate, Hokkaido
  - Novartis Investigative Site, Hakodat, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Sumoto, Hyōgo
  - Novartis Investigative Site, Takarazuka, Hyōgo
  - Novartis Investigative Site, Inashiki, Ibaraki
  - Novartis Investigative Site, Ishioka, Ibaraki
  - Novartis Investigative Site, Mito, Ibaraki
  - Novartis Investigative Site, Kita-gun, Kagawa-ken
  - Novartis Investigative Site, Kagoshima, Kagoshima-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Nankoku, Kochi
  - Novartis Investigative Site, Arao, Kumamoto
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Yokkaichi, Mie-ken
  - Novartis Investigative Site, Miyakonojō, Miyazaki
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Ueda, Nagano
  - Novartis Investigative Site, Nagasaki, Nagasaki
  - Novartis Investigative Site, Kashihara, Nara
  - Novartis Investigative Site, Jōetsu, Niigata
  - Novartis Investigative Site, Sanjō, Niigata
  - Novartis Investigative Site, Ōita, Oita Prefecture
  - Novartis Investigative Site, Yufu, Oita Prefecture
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Hirakata, Osaka
  - Novartis Investigative Site, Moriguchi, Osaka
  - Novartis Investigative Site, Osaka, Osaka
  - Novartis Investigative Site, Ōsaka-sayama, Osaka
  - Novartis Investigative Site, Sakai, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Iruma-gun, Saitama
  - Novartis Investigative Site, Ohtsu, Shiga
  - Novartis Investigative Site, Oda, Shimane
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Chiyoda-ku, Tokyo
  - Novartis Investigative Site, Edogawa City, Tokyo
  - Novartis Investigative Site, Hachiōji, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Katsushika-ku, Tokyo
  - Novartis Investigative Site, Musashino, Tokyo
  - Novartis Investigative Site, Taito-ku, Tokyo
  - Novartis Investigative Site, Toyama, Toyama
  - Novartis Investigative Site, Akita
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Okayama
  - Novartis Investigative Site, Osaka

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CRTH258B1401 that is getting linked from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18311